CLINICAL TRIAL: NCT00232947
Title: A Non-Inferiority Comparison of Fluviral™ Influenza Vaccine to a U.S. Licensed Inactivated Split-Virion Vaccine (Fluzone®) in Adults ≥ 50 Years Old Living in the Community
Brief Title: Study Comparing Immune Response to, and Safety of, Fluviral and Fluzone Influenza Vaccines in Persons 50 y.o. and Over
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ID Biomedical Corporation, Quebec (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: IDB707-108
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2007-01-22 (Estimated); Status verified 2005-10

CONDITIONS: Influenza
Keywords: vaccine; elderly; immunogenicity; safety
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Influenza virus vaccine (Fluviral)
Biological: Influenza virus vaccine (Fluzone)

SUMMARY:
The goal of this study is to determine whether the immune responses induced by Fluviral, the investigational vaccine, are comparable to those induced by Fluzone, which is an influenza vaccine currently licensed in the U.S. The study focuses on persons 50 years old and over. In addition, the study will compare the rate of reactions to the two vaccines, and the general health of persons who receive them over the 42 days after immunization.

DETAILED DESCRIPTION:
Yearly influenza epidemics are responsible for excess hospitalizations and deaths in the elderly population, and also cause lost work and productivity among the healthy, working elderly. Fluviral, a product now licensed in Canada, is being tested to determine whether it is as active in causing immune responses, and as safe as a currently licensed U.S. vaccine in persons 50 y.o. and over.

ELIGIBILITY:
Inclusion Criteria:

* Stable health status
* Access to a consistent means of telephone contact.
* Comprehension of study requirements, availability for study duration
* Availability and ability to attend scheduled visits
* Females post menopausal, sterile or using accepted contraceptive measures
* Competence to provide informed consent

Exclusion Criteria:

* Presence of significant acute or chronic medical or neuropsych. illness
* New medical or surgical treatment w/i 1 month
* Change in medication dose due to uncontrolled symptoms w/i 1 month
* Hospitalization w/i 1 month
* Any unusual risk (for age group) of serious adverse events w/i 1 month
* Any neuropsychiatric condition altering competence for consent
* Any neuropsychiatric condition preventing accurate safety reports
* Febrile illness on day of treatment
* Employment in professions at high risk of influenza transmission
* Residence in a long-term-care facility or with an immunocompromised person
* Systolic BP over 150, diastolic over 90, resting pulse under 50 or over 100
* Cancer w/i 3 years
* Immunosuppressive of immunodeficient conditions
* Treatment with systemic glucocorticoids > replacement
* Treatment with cytotoxic or immunosuppressant drugs
* Treatment with immune globulins
* Clotting disorders that increase the risks of intramuscular injections
* History of demyelinating disease or GBS
* Pregnancy or nursing
* Absence of contraceptive practices in women with childbearing potential
* Planned administration of non-influenza vaccines within 30 days
* Receipt of any investigational drug within 30 days
* Receipt of immune globulin treatment within 3 months
* Known or suspected allergy to egg proteins, gelatin, or thimerosal
* History of severe adverse reactions toflu vaccines
* Prior receipt of 2005-6 influenza vaccine

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900
Dates: Start 2005-10; Study Completion 2006-02

PRIMARY OUTCOMES:
Rate of signficant rises in serum antibody titers against viruses in the vaccines.
Geometric mean serum antibody titers on day 21.

SECONDARY OUTCOMES:
Rates of specific, solicited vaccine reactogenicicty complaints.
Rates of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bouveret, MD, Study Director — ID Biomedical of Quebec
Locations (10):
- United States (10):
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Radiant Research, Atlanta, Georgia
  - Radiant Research, Chicago, Illinois
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - Regional Clinical Research, Endwell, New York
  - University of Rochester Medical Center, Rochester, New York
  - Radiant Research, Cincinnati, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - PI-Coor Clinical Research, Fairfax, Virginia